CLINICAL TRIAL: NCT02838667
Title: Prevention and Early Detection and Intervention of Post-Coronary Artery Bypass Grafting Surgery (CABG) Acute Kidney Injury (AKI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Qi Qian, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-003845
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Acute Renal Injury; Preventive Measures
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): If participants are randomized into the non-intervention group, the participants' information during the study period will be collected. Participants will be managed by a care provider as per the standard of care. Participants may receive nephrology consultation as indicated clinically.
- Standard of Care plus Nephrology Care (Experimental): If participants are randomized into the intervention group, participants' information will be checked by the study investigators daily for 7 days (2 days pre-op and 5 days post-op). When appropriate, investigators may give suggestions to minimize the participants' risk(s) for AKI. Participant's primary care providers may take the suggestions into consideration. Participants' primary care providers are not obligated to carry out the suggestions that are given.
  Interventions: Procedure: Standard of Care plus Nephrology Care

INTERVENTIONS:
Procedure: Standard of Care plus Nephrology Care
  Arms: Standard of Care plus Nephrology Care

SUMMARY:
Nephrology participation in care of patients undergoing CABG could reduce AKI through correction of modifiable risk factors and early detection and intervention of post-op AKI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age >18 years)
* Elective CABG at Mayo Clinic Rochester and Shanghai Zhongshan Hospital from 7/1/2016 to 6/30/2017

Exclusion Criteria:

* Non-elective CABG
* Renal failure on dialysis
* Renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Perfusion pressures (mean arterial pressure) ≥ 65-70 mmHg | baseline to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Qi Qian, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials